CLINICAL TRIAL: NCT05733598
Title: A Phase 2, Open-label, Multicenter Study Investigating RP2 Oncolytic Immunotherapy in Combination With Second-line Therapy in Patients With Locally Advanced Unresectable, Recurrent and/or Metastatic Hepatocellular Carcinoma
Brief Title: Study of RP2 in Combination With Second-line Therapy in Patients With Locally Advanced or Metastatic HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP2-003
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Biliary Tract Cancer
Keywords: Oncolytic virus; Hepatocellular Carcinoma; HCC; Biliary Tract Cancer; BTC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Biliary Tract Neoplasms | interventions — Bevacizumab; atezolizumab; durvalumab

STUDY DESIGN:
Intervention Model Description: This study will enroll patients with locally advanced unresectable, recurrent, and/or metastatic HCC (second line) and patients with unresectable locally advanced or metastatic BTC (first line after chemotherapy discontinuation). Study periods include Screening (28 days), Treatment, and Follow-Up.
  HCC Cohorts 1a/1b/2: First tumor assessment at Week 10 (±3 days) from first dose; second: 9 (±3 days) weeks later; then every 8 weeks (Q8W).
  BTC Cohort 3: First assessment at Week 8 (±3 days); then Q8W. Safety Follow-Up: 30 and 60 days after last RP2 dose; 135 days after last atezolizumab, bevacizumab, or durvalumab dose.
  Efficacy Follow-Up: Imaging every 12 weeks. Survival Follow-Up: Collected by phone every 3 months for up to 3 years from first RP2 dose or until death.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RP2+Bevacizumab and Atezolizumab (Experimental): HCC Cohort 1a and 1b: Patients with locally advanced unresectable, recurrent and/or metastatic HCC who have progressed on 1 prior systemic treatment, which must have included anti-programmed cell death 1 (PD-1)/anti-PD-L1 therapy. Patients will receive atezolizumab plus bevacizumab therapy combined with RP2.
  In cohort 1a, patients will receive RP2 intratumorally every 2 weeks (Q2W) for 4 doses, then every 3 weeks (Q3W) for 4 doses combined with atezolizumab plus bevacizumab.
  In cohort 1b, patients will receive RP2 intratumorally every 2 weeks (Q2W) for 8 doses combined with atezolizumab plus bevacizumab.
  Interventions: Biological: RP2; Biological: Bevacizumab; Biological: Atezolizumab
- RP2 Monotherapy (Experimental): HCC Cohort 2: Patients with locally advanced unresectable, recurrent and/or metastatic HCC who have progressed on 1 prior systemic treatment, which must have included anti-programmed cell death 1 (PD-1)/anti-PD-L1 therapy. Patients will receive RP2 monotherapy every 2 weeks (Q2W).
  Interventions: Biological: RP2 Monotherapy
- RP2+Durvalumab (Experimental): BTC Cohort (Cohort 3): Patients with locally advanced or metastatic BTC (intrahepatic or extrahepatic cholangiocarcinoma or gall bladder carcinoma), who have received treatment with combination gemcitabine, platinum-containing chemotherapy, and checkpoint inhibitor for a minimum of 12 weeks (4 to 8 cycles) and maximum of 24 weeks, and who have had stable disease or partial response on 2 on treatment scans and no progressive disease. After the last combination chemotherapy treatment, checkpoint inhibitor treatment must be limited to 2 doses (8 weeks). Patients will receive durvalumab combined with RP2.
  Interventions: Biological: RP2; Biological: Durvalumab

INTERVENTIONS:
Biological: RP2 — Genetically modified herpes simplex type 1 virus for tumor lysis and immune stimulation.
  Arms: RP2+Bevacizumab and Atezolizumab; RP2+Durvalumab
Biological: Bevacizumab — Anti-VEGF therapy.
  Other Names: Avastin
  Arms: RP2+Bevacizumab and Atezolizumab
Biological: Atezolizumab — Anti-PD-L1 monoclonal antibody.
  Other Names: Tecentriq
  Arms: RP2+Bevacizumab and Atezolizumab
Biological: Durvalumab — Anti-PD-L1 monoclonal antibody
  Other Names: Imfinzi
  Arms: RP2+Durvalumab
Biological: RP2 Monotherapy — Genetically modified herpes simplex type 1 virus for tumor lysis and immune stimulation.
  Other Names: RP2
  Arms: RP2 Monotherapy

SUMMARY:
The purpose of this study is to assess the efficacy and safety of RP2 in combination with atezolizumab plus bevacizumab (Cohorts 1a and 1b) and RP2 monotherapy (Cohort 2) in the as second line treatment in patients with locally advanced unresectable, recurrent, and/or metastatic HCC and in combination with durvalumab as treatment in patients with unresectable locally advanced or metastatic BTC.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter study evaluating RP2 oncolytic immunotherapy in combination with atezolizumab plus bevacizumab and RP2 monotherapy as second-line treatment in patients with locally advanced unresectable, recurrent, and/or metastatic HCC and in combination with durvalumab as treatment in patients with unresectable locally advanced or metastatic BTC (Cohort 3).

The study periods will consist of Screening, Treatment, and Follow-Up:

* 28-day Screening Period
* Treatment Period

  * HCC Cohorts (Cohort 1a, 1b, and 2): First tumor assessment at 10 weeks (± 3 days) from the date of the first dose of study treatment and second assessment 9 weeks (± 3 days) later; subsequent assessments every 8 weeks (Q8W)
  * BTC cohort (Cohort 3): First tumor assessment at 8 weeks (± 3 days) from the date of the first dose of study treatment; subsequent assessments Q8W
* Safety Follow-Up

  * 30 days and 60 days after the last dose of RP2
  * 135 days after the last doses of atezolizumab and bevacizumab
  * 135 days after the last dose of durvalumab
* Efficacy Follow-Up:

  - HCC and BTC Cohorts: Imaging and tumor assessments every 12 weeks
* Survival Follow-Up

  * Survival information will be collected over the phone every 3 months for up to 3 years from the patient's first RP2 dose or until death, whichever occurs first

ELIGIBILITY:
Key Inclusion Criteria:

I 1. Male or female ≥ 18 years of age. I 2. (HCC only) Has locally advanced unresectable, recurrent, and/or metastatic HCC, with the diagnosis confirmed by histologic or cytologic analysis or clinical features or imaging criteria (using LI-RADS v2018; [Chernyak 2018]) according to the American Association for the Study of Liver Diseases criteria for patients with cirrhosis (Marrero 2018). Sites should select lesions that are either "probable HCC - LIRADS 4" or "definite HCC - LIRADS 5".

I 3. (HCC only) Must have progressed while on first and only systemic therapy, which must have included anti PD-1 or anti-PD-L1 therapy (eg, atezolizumab plus bevacizumab combination, durvalumab plus tremelimumab combination, durvalumab, pembrolizumab, or nivolumab monotherapy or nivolumab in combination with ipilimumab) as their immediate prior treatment regimen.

I 4. (HCC only) Child-Pugh A, determined within 14 days before first study treatment.

I 5. Has at least 1 measurable tumor of ≥ 1 cm in longest diameter (or ≥ 1.5 cm shortest diameter for lymph nodes) as defined by RECIST 1.1.

I 6. Has injectable tumor(s), which alone or in aggregate, total at least 1 cm in diameter.

I 7. Must be willing to consent to provide fresh tumor biopsy sample or archival tumor biopsy sample obtained within 90 days before the first dose of study treatment.

I 8. Has adequate hematologic function, including: White blood cell (WBC) count ≥ 2.0 × 109/L; absolute neutrophil count (ANC) ≥ 1.5 × 109/L (without granulocyte-colony stimulating factor support); platelet count ≥ 75 × 109/L (without transfusion); hemoglobin ≥ 8.5 g/dL (may have received transfusions; however, patient must not be transfusion-dependent).

I 9. Has adequate hepatic function including: total bilirubin ≤ 3.0 × upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 5.0 × ULN.

I 10. Has adequate renal function, defined as serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 30 mL/minute (measured using Cockcroft-Gault formula).

I 11. Serum albumin ≥ 2.8 g/dL. I 12. Prothrombin time (PT) ≤ 1.5 × ULN (or international normalization ratio [INR] ≤ 1.7) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.

I 13. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.

I 14. Female and male patients who meet the following criteria:

1. Female patients are eligible if not pregnant (see IC #15) or breastfeeding and if one of the following applies 1) is a woman of non-childbearing potential (WNCBP) OR 2) is a woman of childbearing potential and must agree to use a highly effective contraception method during the treatment period, and for at least (a) 90 days after the last dose of RP2 or (b) 5 months after the last dose of atezolizumab, or (c) 6 months after the last dose of bevacizumab, or (d) 90 days after the last dose of durvalumab, whichever is longer.
2. Male patients are eligible to participate if they agree to the following during the study treatment period, and for at least 90 days after the last dose of RP2: refrain from donating fresh unwashed sperm plus either be abstinent from intercourse where pregnancy can occur (abstinent on a long term and persistent basis) OR must agree to use an external condom and also should advise their partner to use a highly effective method of contraception as a condom may break or leak.

I 15. Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) test with a minimum sensitivity of 25 IU/L or equivalent units of β hCG within 72 hours before the first dose and a negative urine pregnancy test on Dose 1 Day 1.

I 16. Capable of giving signed informed consent which includes willingness to comply with the requirements and restrictions listed in the informed consent form and in this protocol.

I 17. (BTC only) Histologically confirmed, unresectable locally advanced or metastatic adenocarcinoma of biliary tract, including cholangiocarcinoma (intrahepatic or extrahepatic) and gallbladder carcinoma whose disease has not progressed following the concurrent treatment with gemcitabine, platinum containing chemotherapy, and checkpoint inhibitors.

Patients must be on combination treatment with gemcitabine, platinum containing chemotherapy, and a checkpoint inhibitor for a minimum of 12 weeksand maximum of 24 weeks. After the last combination chemotherapy treatment (gemcitabine plus platinum chemotherapy), checkpoint inhibitor treatment must be limited to 2 doses (8 weeks).

Note: Patients who develop toxicity and discontinue platinum containing chemotherapy per treating physicians may enroll into the trial as long as they receive gemcitabine and durvalumab for 12 weeks. SD or PR must be documented on at least 2 scans while on prior combination treatment; the second scan can be the same as the baseline scan.

Key Exclusion Criteria:

E 1. (HCC only) Child-Pugh B or C. E 2. (HCC only) Patients with untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding.

Note: Note: All patients in Cohort 1a and 1b must undergo an esophagogastroduodenoscopy (EGD), and all varices (irrespective of size) must be assessed and treated regardless of grade before enrollment. Patients who have undergone endoscopic treatment of all known varices 90 days before initiation of study treatment do not need to repeat the procedure.

Note: EGD is not required for patients in Cohort 2 (RP2 monotherapy). E 3. Significant bleeding event within the last 12 months that places the patient at unjustifiable risk for bleeding from intratumoral injection procedures, based on Investigator or interventional radiologist assessment.

E 4. (HCC only) Macroscopic intravascular invasion into the hepatic and/or portal vein(s) (ie, no Vp4), , vena cava, and/or other major blood vessel, or into the common bile duct(s).

E 5. (HCC only) Histologic evidence of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma with HCC, or other rare HCC variants.

E 6. History of medically refractory hepatic encephalopathy and/or hepato-renal syndrome.

E 7. Disease that is amenable to curative surgical and/or locoregional therapies.

E 8. Presence of liver tumors that are estimated to invade more than one-third of the liver.

E 9. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring drainage within 7 days before enrollment.

E 10. Hepatitis B virus (HBV) DNA > 500 IU/mL obtained within 28 days prior to initiation of study treatment. Co-infection of HBV and hepatitis C virus (HCV) is not allowed.

Note: Patients with HBV DNA ≤ 500 U/mL are eligible to enroll in the study. Patients must be on anti-HBV treatment (per local standard care that do not have activity with HSV. Entecavir, tenofovir, telbivudine, lamivudine can be used. Anti-HBV treatment must be given for a minimum of 14 days prior to Week 1 Day 1 and must continue antiviral treatment for the length of the study.

E 11. Known human immunodeficiency virus (HIV) infection. Note: Testing for HIV is not required unless mandated by local health authority or clinically indicated.

E 12. Active significant herpetic infections or prior complications of HSV-1 infection (eg, herpetic keratitis or encephalitis) or requires intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).

Note: Patients with sporadic cold sores may be enrolled if no active cold sores are present at the time of Dose 1 Day 1.

E 13. Systemic infection requiring IV antibiotics or other serious infection within 14 days before dosing.

E 14. Received a live vaccine within 28 days before the first dose of study treatment.

E 15. Known central nervous system (CNS) metastases and/or carcinomatous meningitis.

E 16. Prior malignancy, other than HCC and BTC, active within the previous 3 years, except for localized cancers that have apparently been cured or only required surveillance (eg. basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast).

E 17. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study treatment.

Note: Patients who have entered the follow-up phase of an investigational study may participate if it has been 4 weeks after the last dose of the previous investigational agent.

E 18. Systemic anticancer therapies within 4 weeks of the first dose of study drug.

Note: Patients must have recovered (to Grade ≤ 1 or baseline) from all AEs due to previous therapies. Patients with Grade ≤ 2 neuropathy may be eligible if approved by the Medical Monitor.

E 19. Received radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities (except for radiation-induced xerostomia), not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-CNS disease.

E 20. Received prior treatment with an oncolytic virus therapy. E 21. History of significant cardiac disease including myocarditis or congestive heart failure (defined as New York Heart Association Functional Classification III or IV), or unstable angina, serious uncontrolled cardiac arrhythmia, or myocardial infarction within 6 months of enrollment.

E 22. Uncontrolled infection requiring intravenous antibiotics. E 23. History of interstitial lung disease, idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), non-infectious pneumonitis that required steroids, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

E 24. Active tuberculosis. E 25. History or evidence of psychiatric, substance abuse, or any other clinically significant disorder, condition, or disease (except for those outlined above) that, in the opinion of the Investigator or the Medical Monitor, would pose a risk to patient safety or interfere with the study evaluation, procedures, or completion.

E 26. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

E 27. Active, known, or suspected autoimmune disease requiring systemic treatment.

Note: Patients with type 1 diabetes mellitus and/or hypothyroidism requiring only hormone replacement, and/or with autoimmune skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, and/or prior non-serious autoimmune conditions not expected to recur are permitted to enroll.

E 28. Conditions requiring treatment with immunosuppressive doses (> 10 mg per day of prednisone or equivalent) of systemic corticosteroids within 14 days before Dose 1 Day 1.

Note: Patients who require a brief course (≤ 7 days) of corticosteroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. Physiologic replacement doses of systemic corticosteroids are permitted, only if the dose does not exceed 10 mg/day prednisone equivalent.

E 29. Sensitivity to any of the study interventions, or components or thereof, or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

E 30. History of life-threatening toxicity related to prior immune therapy (eg, anti-cytotoxic T lymphocyte antigen 4 or anti-PD-1/anti-PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways [eg, CD40, 4 1BB]) except those that are unlikely to recur or are expected to be manageable with standard countermeasures (eg, hormone replacement after adrenal crisis). Individual cases should be discussed with Medical Monitor if needed.

E 31. (HCC only) Current or recent (within 10 days of first dose of study treatment) use of aspirin or treatment with dipyridamole, ticlopidine, clopidogrel, or cilostazol. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose.

Note: Prophylactic anticoagulation for the patency of venous access devices is allowed.

E 32. Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks before treatment.

E 33. Prior organ transplantation including allogeneic stem-cell transplantation.

E 34. (HCC only) Major surgery within 28 days before starting bevacizumab or anticipated major surgery while on study.

Note: If a patient received major surgery, they must have recovered adequately from the intervention before starting study treatment and must have adequate wound healing, based on Investigator's assessment or surgeon's assessment, before starting bevacizumab.

E 35. (BTC only) Ampullary carcinoma or mixed cholangiocarcinoma with HCC. E 36. (BTC only) Patients with mismatch repair deficiency and microsatellite instability-high are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate per modified RECIST 1.1 | From Day 1 up to 3 years after first RP2 dose of last patient.
  The proportion of patients achieving a BOR of CR or PR per RECIST 1.1 among those that are evaluable for response.

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) | From Day 1 up to 135 days after last dose.
  The incidence of all TEAEs
ORR per RECIST modified for HCC (HCC mRECIST) for HCC cohort only | From Day 1 up to 3 years after first RP2 dose of last patient
  The proportion of patients achieving a BOR of CR or PR per HCC-mRECIST among those that are evaluable for response
Duration of response (DOR) | From Day 1 up to 3 years after first RP2 dose of last patient.
  The time from a tumor response, either a CR or PR (whichever is recorded first), until the date of PD, which was subsequently confirmed, or with no further follow up, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: May Cho, MD, Study Director — Replimune Inc.
Locations (11):
- United States (11):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Sylvester Comprehensive Cancer Center (University of Miami Hospital and Clinics), Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Montefiore Medical CenterMontefiore Medical Park, The Bronx, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The West Clinic, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee